CLINICAL TRIAL: NCT03962608
Title: Safety and Tolerability of Yaq-001 in Patients With Non-Alcoholic Steatohepatitis ("NASH-Safety")
Brief Title: Safety and Tolerability of Yaq-001 in Patients With Non-Alcoholic Steatohepatitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not approved by Health Authorities until get the results of the previous study
Sponsor: Yaqrit Ltd (Industry)
Collaborators: University College, London (Other); Servicio Madrileño de Salud, Madrid, Spain (Other); Hospital Universitari Vall d'Hebron Research Institute (Other); Azienda Ospedaliera di Padova (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); University of Bern (Other); Assistance Publique - Hôpitaux de Paris (Other); University of Lisbon (Other); Alpha Bioresearch S.L. (Other); Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); University of Brighton (Other); A2F Associates Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Yaq001-S-002
Record Dates: First submitted 2019-05-15; First posted 2019-05-24 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Non-Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Randomized (1:1) to:
  * Standard medical treatment + Yaq-001 (8 g/ day) - n= 35
  * Standard medical treatment + placebo-control (placebo for 8 g of Yaq-001/ day) - n= 35
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yaq-001 (Experimental): Standard medical treatment + Yaq-001 (8 g/ day)
  Interventions: Device: Yaq-001
- Placebo (Placebo Comparator): Standard medical treatment + placebo-control (placebo for 8 g of Yaq-001/ day)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Yaq-001 — Study patients will be dosed daily with 8g of product Yaq-001 for a period of 48 weeks. The product will be provided as beads packed in individual sachets intended each for one oral administration. For each patient, the study duration will be up to 54 weeks, including the screening (up to 45 days), treatment (48 weeks) and 7-day follow up period.
  Arms: Yaq-001
Device: Placebo — Study patients will be dosed daily with a quantity of placebo equivalent to 8g of product Yaq-001 for a period of 48 weeks. The product will be provided as beads packed in individual sachets intended each for one oral administration. For each patient, the study duration will be up to 54 weeks, including the screening (up to 45 days), treatment (48 weeks) and 7-day follow up period.
  Arms: Placebo

SUMMARY:
Gut-derived endotoxaemia, microbial imbalance and bacterial translocation play an increasingly recognized role in the progression from non-alcoholic fatty liver disease (NAFLD) to its more advanced state, NASH (non-alcoholic steatohepatitis). Animal model studies confirmed that Yaq-001 reduces liver injury and prevents steatosis in these models which leads to the theoretical potential of Yaq-001 altering the microbiome and gut permeability in patients with NASH.

The purpose of this clinical trial is to study the safety and tolerability of Yaq-001 in patients with NASH. Results from this study will lead to the design of future pivotal performance and safety trials for registration purposes.

Candidate patients must be between 18-70 years old and have a clinical diagnosis of NASH, determined histologically or phenotypically, as well as meeting other clinical inclusion/exclusion criteria.

Eligible patients will be randomly assigned to receive standard of care treatment plus Yaq-001, or standard of care treatment plus placebo).

The treatment lasts for 48 weeks. During treatment, the patient will have 6 study visits. At all the visits, the patients will undergo a routine physical examination, electrocardiogram, collection of blood and urine samples. On three occasions the patients will be asked to provide additional samples of blood, urine and stool for analysis outside the hospital. On two occasions the patient will have a liver Multiscan and on three occasions the patient will have a liver Fibroscan.

70 patients from 9 hospitals in UK, France, Italy, Portugal, Spain and Switzerland will participate in this study.

DETAILED DESCRIPTION:
This is a multicentre, randomized, double blinded, placebo controlled trial to intended to evaluate safety and tolerability of oral administration of Yaq-001 therapy.

70 Non-Alcoholic Steatohepatitis patients will be randomized (1:1) to:

* Standard medical treatment + Yaq-001 (8 g/ day) - n= 35
* Standard medical treatment + placebo-control (placebo for 8 g of Yaq-001/ day) - n= 35

Study patients will be dosed daily with Yaq-001 (or an equivalent quantity of placebo) for 48 weeks.

Assessment of DSMB will take place when 15 Yaq-001- and 15 placebo-treated patients have completed 12 weeks of dosing.

Investigational centres specialized in the management of patients with Non-Alcoholic Steatohepatitis will participate in the study.

For each patient, the study duration will be up to 54 weeks, including the screening (up to 45 days), treatment (48 weeks) and 7-day follow up period.

The total study duration is estimated to be approximately 18 months from screening of first patient until study completion of the last patient.

This project has received funding from the European Union's Horizon 2020 research and innovation programme.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 <70 years at screening
2. HbA1C < 10.5%
3. BMI >25kg/m2
4. ALT <250IU/L
5. Ability to provide informed consent
6. Agree to the use of effective contraceptive measures if either male or female of child bearing potential.

Exclusion Criteria:

1. History of metabolic acidosis or ketoacidosis
2. Presence of vascular liver disease
3. Cirrhosis diagnosed either histologically, by laboratory or clinically;
4. Presence of liver disease of other aetiology (autoimmune, metabolic, medication induced);
5. HIV antibody positive, hepatitis B surface antigen positive (HBsAg) or Hepatitis C virus (HCV)-RNA positive;
6. Current or history of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to screening (significant alcohol consumption is defined as more than 20 grams per day in females and more than 30 grams per day in males, on average)
7. Type 1 diabetes;
8. History of bariatric intervention (surgical or endoscopic) performed 6 months or more prior to screening;
9. Weight loss or gain of 5kg or more in the past 3 months or >10% change in bodyweight in the past 3 months;
10. Inadequate venous access;
11. Lactating/breastfeeding/pregnant at Screening or Baseline;
12. Receiving an elemental diet or parenteral nutrition;
13. Medical conditions, such as:

    * Inflammatory bowel disease;
    * Unstable angina, myocardial infarction, transient ischemic events, or stroke within 24 weeks of Screening;
    * Active infection
    * Active autoimmune disease
    * Malignant disease at any time
    * Severe congestive heart failure (current medical therapy or current clinical evidence of congestive heart failure NHYA class III/IV) Persistent, uncontrolled hypertension despite optimal medical treatment (for example: Systolic blood pressure (SBP) >160 mmHg or diastolic blood pressure (DBP) >100 mmHg (average of 2 readings) measured in the sitting position at Visit 1, after at least 5 minutes seated rest at screening).
    * Any other medical condition which, in the opinion of the investigator, could impact adversely on the subject participating or on the interpretation of the study data
    * Presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, metabolic, haematological, neurological, psychiatric, systemic, ocular, gynaecologic or any acute infectious disease or signs of acute illness that, in the opinion of the investigator, might compromise the patient's safe participation in the trial
14. Concurrent medications including:

    * Anti-NASH therapy(s) taken for more than 10 continuous days in the last 3 months. These include S-adenosyl methionine (SAM-e), betaine, milk thistle, probiotic supplements (other than yoghurt), vitamin E and gemfibrozil.
    * Wash out for any of the anti-NASH therapies is as follows: under 10 days no washout required, more than 10 days and up to 3 months treatment requires 6 weeks washout.
    * Use of drugs historically associated with non-alcoholic fatty liver disease (NAFLD) (amiodarone, methotrexate, systemic glucocorticoids, tetracyclines, tamoxifen, estrogens at doses greater than those used for hormone replacement, anabolic steroids, valproic acid, and other known hepatotoxins) during the previous year prior to randomization
    * Thiazolidinediones (glitazones), or glucagon-like peptide-1 analogues in the last 90 days.

      1. NOTE: Allowable anti-diabetic treatment includes metformin and/or sulfonylureas and/or dipeptidyl peptidase 4 inhibitors (gliptins) administered at constant dose for at least 2 months prior to study entry
      2. NOTE: Subjects treated with Insulin are eligible if clinically stable on insulin treatment (i.e. no recurrent acute hypo-/hyperglycaemic episodes diagnosed clinically and by Glucose serum levels of <50 mg/dL and >200 mg/dL respectively) for at least 2 months prior to study entry
    * immune modulatory agents including: systemic steroids for more than 7 days; daily treatment with multiple non-steroidal anti-inflammatory drugs (such as aspirin (>100mg/day), ibuprofen, naproxen, meloxicam, celecoxib) for more than 1 month
    * Use of ursodeoxycholic acid (Ursodiol, Urso) or obeticholic acid (Ocaliva) within 90 days prior to enrolment

    In the last 6 months:
    * azathioprine, 6-mercaptopurine, methotrexate, cyclosporin, anti-TNFα therapies (infliximab, adalimumab, etanercept) or anti-integrin therapies (namixilab)
    * More than 10 consecutive days oral or parenteral antibiotics within 4 weeks prior to study entry. NOTE: subjects administered with antibiotics for more the 5 days prior to study entry would not be included in the stool and PBMC analysis

    Within the preceding 4 weeks before treatment:

    - immunosuppression, long acting benzodiazepine or barbiturates and antiviral medication
15. The following laboratory abnormalities:

    * Neutrophil count ≤1.0 x 109/L; Platelets <100 x 109/L
    * Haemoglobin <10g/dL; Albumin <3.5g/dL
    * International Normalized Ratio (INR) >1.5
    * Total bilirubin >1.5 x upper limit of reference range (unless Gilbert's syndrome or extrahepatic source as denoted by increased indirect bilirubin fraction)
    * Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2 at Screening or Baseline using the Modification of Diet in Renal Disease (MDRD) equation.
    * Creatine Phosphokinase >5x ULN
16. Past history of acute pancreatitis with current triglycerides 400 mg/dL at Visit 1.
17. Any planned major surgery to be performed during the study (e.g., coronary artery bypass surgery, abdominal aortic aneurysm repair, etc.).
18. Clinical evidence of hepatic decompensation as defined by the presence of any of the following abnormalities:

    * Serum albumin less than 3.4 grams/deciliter (g/dL)
    * International Normalized Ratio (INR) greater than 1.3
    * Total bilirubin greater than 1.5 milligrams per deciliter (mg/dL)
    * Direct bilirubin greater than 0.4 milligrams per deciliter (mg/dL)
    * History of esophageal varices, ascites or hepatic encephalopathy
19. Evidence of other forms of chronic liver disease:

    * Hepatitis B as defined by presence of hepatitis B surface antigen (HBsAg)
    * Hepatitis C as defined by presence of hepatitis C virus (HCV) ribonucleic acid (RNA) within last two years.
    * Evidence of ongoing autoimmune liver disease as defined by compatible liver histology
    * Primary biliary cirrhosis as defined by the presence of at least 2 of these criteria (i) Biochemical evidence of cholestasis based mainly on alkaline phosphatase elevation (ii)Presence of anti-mitochondrial antibody (AMA) (iii)Histologic evidence of non-suppurative destructive cholangitis and destruction of interlobular bile ducts
20. Serum creatinine of ≥2.0 mg/dL
21. History of biliary diversion
22. Participation in any clinical study of an investigational medicinal product within 30 days or five half-lives of the investigational product, whichever is longer.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-31 (Estimated); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of reported and observed Serious Adverse Events | Day 1
  The percentage of patients experiencing SAEs will be tabulated by arm.
Assessment of reported and observed Serious Adverse Events | Week 1
  The percentage of patients experiencing SAEs will be tabulated by arm.
Assessment of reported and observed Serious Adverse Events | Week 12
  The percentage of patients experiencing SAEs will be tabulated by arm.
Assessment of reported and observed Serious Adverse Events | Week 24
  The percentage of patients experiencing SAEs will be tabulated by arm.
Assessment of reported and observed Serious Adverse Events | Week 36
  The percentage of patients experiencing SAEs will be tabulated by arm.
Assessment of reported and observed Serious Adverse Events | Week 48
  The percentage of patients experiencing SAEs will be tabulated by arm.
Assessment of treatment-related Serious Adverse Events | Day 1
  The percentage of patients experiencing device-related SAEs will be tabulated by arm.
Assessment of treatment-related Serious Adverse Events | Week 1
  The percentage of patients experiencing device-related SAEs will be tabulated by arm.
Assessment of treatment-related Serious Adverse Events | Week 12
  The percentage of patients experiencing device-related SAEs will be tabulated by arm.
Assessment of treatment-related Serious Adverse Events | Week 24
  The percentage of patients experiencing device-related SAEs will be tabulated by arm.
Assessment of treatment-related Serious Adverse Events | Week 36
  The percentage of patients experiencing device-related SAEs will be tabulated by arm.
Assessment of treatment-related Serious Adverse Events | Week 48
  The percentage of patients experiencing device-related SAEs will be tabulated by arm.
Assessment of withdrawals due to Adverse Events | Day 1
  The percentage of patients who withdraw due to an AE will be tabulated by arm.
Assessment of withdrawals due to Adverse Events | Week 1
  The percentage of patients who withdraw due to an AE will be tabulated by arm.
Assessment of withdrawals due to Adverse Events | Week 12
  The percentage of patients who withdraw due to an AE will be tabulated by arm.
Assessment of withdrawals due to Adverse Events | Week 24
  The percentage of patients who withdraw due to an AE will be tabulated by arm.
Assessment of withdrawals due to Adverse Events | Week 36
  The percentage of patients who withdraw due to an AE will be tabulated by arm.
Assessment of withdrawals due to Adverse Events | Week 48
  The percentage of patients who withdraw due to an AE will be tabulated by arm.

SECONDARY OUTCOMES:
Determine potential of Yaq-001 for the treatment of NASH | From Baseline at 48 Weeks
  Mean change in alterations in hepatic fat fraction (steatosis) as evaluated by MRI -PDFF
Determine potential of Yaq-001 for the treatment of NASH | From Baseline at 48 Weeks
  Mean change in alterations in fibrosis as evaluated by corrected LMS T1 score
Determine potential of Yaq-001 for the treatment of NASH | From Baseline at 24 and 48 weeks
  Mean change in alterations in median stiffness as determined by Fibro-scanning
Determine potential of Yaq-001 for the treatment of NASH | From Baseline at 24 and 48 weeks
  Mean change in alterations in enhanced liver fibrosis (ELF) scores as non-invasive markers of liver fibrosis
Determine potential of Yaq-001 for the treatment of NASH | From Baseline at 24 and 48 weeks
  Mean change in alterations in markers of insulin resistance (homeostatic assessment method, HOMA-IR score)
Determine potential of Yaq-001 for the treatment of NASH | From Baseline at 24 and 48 weeks
  Mean change in alterations in glucose levels
Determine potential of Yaq-001 for the treatment of NASH | From Baseline at 24 and 48 weeks
  Mean change in changes in the levels of glycated haemoglobin (HbA1C)
Determine potential of Yaq-001 for the treatment of NASH | From Baseline at 24 and 48 weeks
  Analytical to see the mean change in serum lipid profile
Determine potential of Yaq-001 for the treatment of NASH | From Baseline at 24 and 48 weeks
  Change from baseline in serum levels of cytokeratin (CK)18 - M30 and M65 fractions as indicators of hepatocellular apoptosis and necrosis
Determine potential of Yaq-001 for the treatment of NASH | From Baseline at 24 and 48 weeks
  Mean change in microbiome composition
Determine potential of Yaq-001 for the treatment of NASH | From Baseline at 1, 12, 24, 36 and 48 weeks
  Mean change in alterations in the level of the fibrosis-4 (FIB-4)
Determine potential of Yaq-001 for the treatment of NASH | From Baseline at 1, 12, 24, 36 and 48 weeks
  Mean change in alterations in the Non-Alcoholic Fatty liver disease fibrosis (NAFLD-F). Fibrosis will be measured by liver multiscan, fibroscan and serological markers of fibrosis defined in the protocol.
Determine potential of Yaq-001 for the treatment of NASH | From Baseline at 1, 12, 24, 36 and 48 weeks
  Mean change in alterations in liver biochemistry as detected by changes in serum Alanine Aminotransferase (ALT)
Determine potential of Yaq-001 for the treatment of NASH | From Baseline at 1, 12, 24, 36 and 48 weeks
  Mean change in alterations in liver biochemistry as detected by changes in serum Aspartate transaminase (AST)
Determine potential of Yaq-001 for the treatment of NASH | From Baseline at 1, 12, 24, 36 and 48 weeks
  Mean change in alterations in liver biochemistry as detected by changes in serum gamma glutamyl transferase (GGT)
Determine potential of Yaq-001 for the treatment of NASH | From Baseline at 1, 12, 24, 36 and 48 weeks
  Mean change in alterations in liver biochemistry as detected by changes in serum alkaline phosphatase
Determine potential of Yaq-001 for the treatment of NASH | From Baseline at 1, 12, 24, 36 and 48 weeks
  Mean change in alterations in liver biochemistry as detected by changes in serum bilirubin
Assessment of changes in nutritional status | From Baseline at 1, 12, 24, 36, 48 weeks and Termination visit
  Clinical nutritional assessment, (weight and height will be combined to report BMI in kg/m^2)
Assessment of changes in nutritional status | From Screening, Baseline at 1, 12, 24, 36 and 48 weeks
  Laboratory assessment of micronutrients: Local labs: Vitamin B9
Assessment of changes in nutritional status | From Screening, Baseline at 1, 12, 24, 36 and 48 weeks
  Laboratory assessment of micronutrients: Local labs: Vitamin B12
Assessment of changes in nutritional status | From Screening, Baseline at 1, 12, 24, 36 and 48 weeks
  Laboratory assessment of micronutrients: Local labs: Vitamin D
Assessment of changes in nutritional status | Baseline, Weeks 24 and 48
  Laboratory assessment of micronutrients: Core labs (blood): Vitamins B1
Assessment of changes in nutritional status | Baseline, Weeks 24 and 48
  Laboratory assessment of micronutrients: Core labs (blood): Vitamins B2
Assessment of changes in nutritional status | Baseline, Weeks 24 and 48
  Laboratory assessment of micronutrients: Core labs (blood): Vitamins B3
Assessment of changes in nutritional status | Baseline, Weeks 24 and 48
  Laboratory assessment of micronutrients: Core labs (blood): Vitamins A
Assessment of changes in nutritional status | Baseline, Weeks 24 and 48
  Laboratory assessment of micronutrients: Core labs (blood): Vitamins E
Assessment of changes in nutritional status | Baseline, Weeks 24 and 48
  Laboratory assessment of micronutrients: Core labs (blood): Vitamins K
Assessment of changes in nutritional status | Baseline, Weeks 24 and 48
  Laboratory assessment of micronutrients: Core labs (blood): zinc (Zn)
Assessment of changes in nutritional status | Baseline, Weeks 24 and 48
  Laboratory assessment of micronutrients: Core labs (blood): Copper (Cu)
Assessment of changes in nutritional status | Baseline, Weeks 24 and 48
  Laboratory assessment of micronutrients: Core labs (blood): Selenium (Se)
Assessment of changes in nutritional status | Baseline, Weeks 24 and 48
  Laboratory assessment of micronutrients: Core labs (urine): niacin metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Jalan, Study Chair — Head, Liver Failure Group ILDH, Division of Medicine UCL Medical School Royal Free Campus Rowland Hill Street London NW32PF; Jane Macnaughtan, Study Director — Consultant, Liver Failure Group, ILDH, Division of Medicine UCL Medical School Royal Free Campus Rowland Hill Street London NW32PF
Locations (9):
- Hospital Beaujon, Hepatology and Liver Intensive Care,, Clichy, France
- Italy (2):
  - Policlinico S.Orsola Malpighi, Department of Medical and Surgical Sciences, Bologna
  - Azienda Ospedaliera di Padova, Hepatic Emergencies Unit, Padua
- University Hospital of Santa Maria, Lisbon, Portugal
- Spain (3):
  - Hospital Vall d'Hebron, Liver Unit, Barcelona
  - Hospital Clinic of Barcelona , Liver Unit,, Barcelona
  - Hospital Ramon y Cajal, Department of Gastroenterology and Hepatology, Madrid
- Inselspital Universitaet Bern, Department for Visceral Surgery and Medicine, Bern, Switzerland
- Royal Free Hospital, Institute of Liver and Digestive Disease, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No